CLINICAL TRIAL: NCT04394455
Title: Effect of Brief Cognitive Behavioral Therapy Versus Crisis Intervention Therapy Through Telepsychiatry in Medical Staff During the COVID-19 Pandemic: A Multicentric Randomized Controlled Trial
Brief Title: Brief Cognitive Behavioral Therapy Versus Crisis Intervention Therapy Through Telepsychiatry on Psychiatric Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Principal Investigator, Hector Benjamin Valle Rodriguez, Chief Resident, Universidad Nacional Autonoma de Honduras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1503202018052020242912
Record Dates: First submitted 2020-05-03; First posted 2020-05-19 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Anxiety; Depressive Symptoms; Post Traumatic Stress Symptoms; Perceived Stress
Keywords: telepsychiatry; cognitive behavioral therapy; crisis intervention; anxiety; depression; post traumatic stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The interventional models are brief cognitive behavioral therapy and crisis intervention therapy through telepsychiatry. Each arm will be divided into therapy groups with a maximum of 10 participants per group. Each therapy session will be directed by a therapist and a co-therapist using a predefined structure for each intervention, with a duration of 60-90 minutes per session.
Who Masked: Investigator
Masking Description: Investigators will not take part in the baseline symptom evaluation of subjects or the post-intervention evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief cognitive behavioral therapy (Experimental): Medical staff (medical doctors and residents) who will receive brief cognitive behavioral therapy through telepsychiatry.
  Interventions: Behavioral: Brief cognitive behavioral therapy
- Crisis intervention therapy (Active Comparator): Medical staff (medical doctors and residents) who will receive 3 sessions of crisis intervention therapy through telepsychiatry.
  Interventions: Behavioral: Crisis intervention therapy

INTERVENTIONS:
Behavioral: Brief cognitive behavioral therapy — 9 structured psychotherapy sessions, weekly, 60-90 minutes duration. Provided by one therapist and one co-therapist. Provided through telepsychiatry.
  Arms: Brief cognitive behavioral therapy
Behavioral: Crisis intervention therapy — 3 structured sessions of crisis intervention. One session each week for three weeks. Provided by one therapist and one co-therapist. Provided through telepsychiatry.
  Arms: Crisis intervention therapy

SUMMARY:
The purpose of this randomized controlled trial is to determine the effect of two behavioral interventions: brief cognitive-behavioral therapy and crisis intervention therapy through telepsychiatry, over the level of perceived stress, anxiety, depression and post-traumatic stress symptoms during the COVID-19 pandemic in medical residents and medical staff at three hospitals in two cities of Honduras.

DETAILED DESCRIPTION:
The psychotherapeutic interventions are going to be delivered from June to August at each participating center. Subjects will be allocated randomly in each of the two interventional arms independently by stratification in each participating center. The population for intervention will be medical staff from three different national hospitals in the frontline during the pandemic. After valid informed consent, a screening process will take place to identify symptoms as baseline evaluation using validated self-assessment tools delivered through electronic invitation. Post-intervention measurements will take place at 3 and 6 months from baseline. Intention to treat analysis and per-protocol analysis will take place. CONSORT guidelines were followed.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors and medical residents 18 years and older, from UNAH medical school and Hospital de Occidente.
* Medical doctors and medical residents whom during the initial screening show positive scores in Patient Health Questionnaire-2 and Generalized Anxiety Disorder scale-2
* Access to internet and an electronic device

Exclusion Criteria:

* Medical doctors and medical residents referring a history of psychiatric disorders
* Medical residents that belong to the Psychiatry Residency Program
* Medical residents and medical doctors that have been diagnosed with COVID-19
* Medical doctors and residents whom during evaluations show severe symptoms of depression, anxiety and post-traumatic stress symptoms
* Medical doctors and residents with negative screening in Patient Health Questionnaire-2 and Generalized Anxiety Disorder Scale-2
* Participants that do not have access to internet connection or an electronic device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate reduction in Depressive symptoms | 6 months after psychotherapeutic intervention has started
  Patient Health Questionnaire 9 scale (PHQ-9), a 9 item scale with a score range from 0 to 27. A higher score means a worse outcome.
Rate reduction in Anxiety symptoms | 6 months after psychotherapeutic intervention has started
  General Anxiety Disorder 7 Scale (GAD-7), a 7 item scale with a score range from 0 to 21. A higher score means a worse outcome.
Rate reduction in Post traumatic Stress symptoms | 6 months after psychotherapeutic intervention has started
  Post-traumatic Stress Scale for DSM-5 (PCL-5), a 20 item scale with a score range from 0 to 80. A higher score means a worse outcome.
Rate reduction in Perceived stress level | 6 months after psychotherapeutic intervention has started
  Perceived stress scale (PSS), a 10 item scale with a score range from 0 to 40. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: José R Galindo-Donaire, MD, Principal Investigator — Universidad Nacional Autonoma de Honduras; Elena N Reyes-Flores, MD, Principal Investigator — Universidad Nacional Autonoma de Honduras
Locations (1):
- Universidad Nacional Autónoma de Honduras, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No